CLINICAL TRIAL: NCT03777683
Title: Evaluation the Effects of French Maritime Pine Bark Extract Supplementation on the Inflammatory Biomarkers, Nutritional and Clinical Status in Traumatic Brain Injury Patients, in Intensive Care Unit; A Randomized Clinical Trial
Brief Title: Evaluation the Effects of French Maritime Pine Bark Extract on the Clinical Status in Traumatic Brain Injury Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mahsa Malekahmadi, principal investigator, Mashhad University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 970612
Record Dates: First submitted 2018-12-12; First posted 2018-12-17 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Dietary Supplements; Oligopin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: On enrolment, study nutritionist or clinicians take a consecutive sealed opaque envelope containing the unique patient identifier but not the study group, to which they remain masked. A paired set of sealed envelopes are kept in a locked cabinet in the study laboratory, label with the unique patient identifier and containing the study group allocation. These are opened by the nutritionist. Investigators, all study staff hospital attending clinical teams, and patients were masked to the study group allocation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary Supplement (OLIGOPIN) (Experimental): Intervention group will receive French maritime pine bark extract supplement (OLIGOPIN) in the form oral capsules containing 50 mg French maritime pine bark extract plus 130 mg Microcrystalline Cellulose. OLIGOPIN powder of each capsule are dissolved in 10 ml deionized water and given to patients via gavage (3 capsule per day) for 10 days
  Interventions: Dietary Supplement: Dietary Supplement (OLIGOPIN)
- Placebo (Placebo Comparator): Control group will receive oral capsules containing 130 mg Microcrystalline Cellulose with 10 ml of deionized water via gavage (3 capsule per day) for 10 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Dietary Supplement (OLIGOPIN) — investigators obtained ethical approval from the Research Ethics Committees of the Mashhad University of medical sciences. investigators enroll 60 patients who are admitted to ICU at hospitals of university. All eligible patients or their first degree relatives give informed consent before participating. Participants are randomly (block stratification) divided in two groups. At the first visit, baseline data are gathered and intervention group (n=30) will receive Oligopin supplement. In order to control the confounding effect of food intake, both the control and the intervention group receive the standard formulas based on their daily required energy via enteral root feeding.
  Arms: Dietary Supplement (OLIGOPIN)
Other: Placebo — investigators obtained ethical approval from the Research Ethics Committees of the Mashhad University of medical sciences. investigators enroll 60 patients who are admitted to ICU at hospitals of university. All eligible patients or their first degree relatives give informed consent before participating. Participants are randomly (block stratification) divided in two groups. At the first visit, baseline data are gathered and control group (n=30) will receive oral capsules containing 130 mg Microcrystalline Cellulose. In order to control the confounding effect of food intake, both the control and the intervention group receive the standard formulas based on their daily required energy via enteral root feeding.
  Arms: Placebo

SUMMARY:
Introduction: Traumatic brain injury (TBI) is one of the major health and socioeconomic problems in the world. Immune-enhancing enteral formula has been proven to significantly reduce infection rate in TBI patient. One of the ingredients that can be used in immunonutrition formulas to reduce inflammation and oxidative stress is French maritime pine bark extract.

Objective: The main objective of present study is surveying the effect of French maritime pine bark extract on the clinical, nutritional and inflammatory status of TBI patients as the first human study in the world.

Method: this is double-blind, randomized controlled trial. Block randomization are used. Intervention group will receive French maritime pine bark extract supplement (OLIGOPIN) 150 mg for 10 days. Control group will receive placebo for the same duration. Inflammatory status (IL-6, IL- 1β, C-reactive protein) and oxidative stress status (Malondialdehyde, total antioxidant capacity), at the base line, at the 5th day and at the end of the study (10th day) are measured. APACHE ІІ (acute physiologic and chronic health evaluation II) for assessment of clinical status of patients and Nutric questionnaires for assessment of nutritional status filled out at the base line, 5th day and the end of study. SOFA (sequential organ failure assessment) questionnaire for assessment of organ failure filled out every other day. The mortality rate will be asked by phone within 28 days of the start of the intervention. Weight, body mass index and body composition at baseline, 5th day and 10th day of intervention are measured. All analyses will be conducted by initially assigned study arm in an intention-to-treat analysis. The data will be expressed as mean ± SD.

DETAILED DESCRIPTION:
Randomization:

investigators randomly assign eligible patients on enrolment (1:1) to either the control group or the intervention group. Randomization is stratified by site and a randomization list of unique patient identifiers is generated by the study statistician using a computer-generated random block size. The classification is based on age (18 to 40 and 40 to 65 years old), gender (male / female) and APACHEII score (0 to 35 and 35 to 71) using quadruple blocks.

ELIGIBILITY:
Inclusion Criteria:

* Admission in ICU due to TBI2
* 18 year ≤ age ≤ 65 year
* GCS score ˃ 8
* Stable hemodynamic and metabolic status in the first 24 to 48 hours
* Having enteral nutritional support
* Fill out the informed consent form by the patient or first-degree relatives of the patient

Exclusion Criteria:

* Pregnancy and lactation
* Morbid obesity: BMI ≥ 40
* Failure to start enteral nutrition in the first 24-48 hours
* Suffering from autoimmune disorders and HIV/Aids
* Suffering or having History of cancer and any liver failure
* Receiving positive inotropic medications including Dopamine, Dobutamine and Epinephrine
* Severe and active bleeding
* Suffering from Sepsis
* Having history of known food allergies

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2019-04-14 (Actual); Primary Completion 2019-12-22 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
change of IL-6 | 5 and 10 days
  Inflammatory markers
change of IL-1β | 5 and 10 days
  Inflammatory marker
change of CRP | 5 and 10 days
  Inflammatory marker
change of Malondialdehyde | 5 and 10 days
  Oxidative stress marker
change of total anti- oxidant capacity | 5 and 10 days
  anti-oxidative stress marker
change of weight | 5 and 10 days
  measurement is done via portable scale
change of body fat percentage | 5 and 10 days
  measurement is done via Bio impedance device "Inbody"
change of Body mass index | 5 and 10 days
  it is calculated by Equation
change of acute physiologic and chronic health evaluation II score | 5 and 10 days
  The Acute Physiology and Chronic Health Evaluation (APACHE II) is a severity score and mortality estimation tool developed from a large sample of ICU patients in the United States.
  Interpretation: Score: 0-4: Death Rate (%):4, Score: 5-9:Death Rate (%):8, Score: 10-14:Death Rate (%):15, Score: 15-19:Death Rate (%):25, Score: 20-24:Death Rate (%):40, Score: 25-29:Death Rate (%):55, Score: 30-34:Death Rate (%):75. Score: ˃ 34 :Death Rate (%):85.
change of sequential organ failure assessment score | 1, 3, 5, 7, 9, 10 days
  The Sequential Organ Failure Assessment (SOFA) is a morbidity severity score and mortality estimation tool developed from a large sample of ICU patients throughout the world. The SOFA was designed to focus on organ dysfunction and morbidity, with less of an emphasis on mortality prediction.
  Interpretation: Score: 0-6: Death Rate (%):< 10%, Score: 7-9:Death Rate (%):15 - 20%, Score: 10-12:Death Rate (%):40 - 50%, Score: 13-14:Death Rate (%):50 - 60%, Score: 15:Death Rate (%):> 80%, Score: 15-24:Death Rate (%):> 90%.
change of Nutric score | 5 and 10 days
  The NUTRIC score (Nutrition assessment in critically ill) is a rapid assessment of nutritional state based on illness severity, age and co-morbidities.
  Sum of points: 6-10: CATEGORY: High Score. Sum of points: 0-5: CATEGORY: LOW Score High score associated with worse clinical outcomes (mortality, ventilation).These patients are the most likely to benefit from the aggressive nutrition therapy.
  LOW Score: These patients have a low malnutrition risk

SECONDARY OUTCOMES:
28-day mortality | 28 days
  the rate of mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Mahsa Malekahmadi, Tehran, Iran

REFERENCES:
- [Derived] Malekahmadi M, Moradi Moghaddam O, Islam SMS, Tanha K, Nematy M, Pahlavani N, Firouzi S, Zali MR, Norouzy A. Evaluation of the effects of pycnogenol (French maritime pine bark extract) supplementation on inflammatory biomarkers and nutritional and clinical status in traumatic brain injury patients in an intensive care unit: A randomized clinical trial protocol. Trials. 2020 Feb 11;21(1):162. doi: 10.1186/s13063-019-4008-x. PMID 32046747